CLINICAL TRIAL: NCT04373785
Title: A Multi-Center Pilot/Phase I and Phase II Clinical Trial of NG101m Adjuvant Therapy in Newly Diagnosed Glioblastoma Patients
Brief Title: NG101m Adjuvant Therapy in Glioblastoma Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NeuGATE Theranostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NG101m
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy; Temozolomide

STUDY DESIGN:
Intervention Model Description: Radiation: Radiotherapy Drug: Temozolomide Drug: NG101m
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NG101m and standard treatment (Experimental): Concomittant therapy:
  Radiation therapy, oral temozolomide, and oral NG101m
  Adjuvant therapy:
  Oral temozolomide and oral NG101m
  Interventions: Radiation: Intensity-modulated radiation therapy; Drug: Temozolomide; Drug: NG101m

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy — Intensity-modulated radiation therapy (IMRT) in daily fractions of 2.67 Gy given 5 days per week for 3 weeks, for a total of 40.05 Gy.
  Other Names: radiation therapy
Drug: Temozolomide — Oral temozolomide (75 mg/m2), given 5 days per week, for 3 weeks during radiotherapy.
  1 month after the discontinuation of radiotherapy, oral temozolomide is restarted at 150 to 200 mg/m2 for 5 days during each 28-day cycle for 12 cycles.
  Other Names: Temodar
Drug: NG101m — Oral NG101m capsule continuously twice daily.
  Other Names: NG101m regimen

SUMMARY:
The purpose of this clinical trial is to evaluate the addition of NG101m adjuvant therapy to standard of care treatment of glioblastoma multiforme. All subjects will receive NG101m capsules along with the standard treatment of temozolomide and radiation.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM) is the most lethal form of malignant brain cancer, with about 12,000 new cases diagnosed each in the the United States. The current standard treatment consists of maximal, safe resection, followed by radiation therapy of 60 Gray (Gy) with concomitant oral temozolomide (TMZ) for 6 weeks, then continue with six cycles of high-dose temozolomide. The median survival rate for newly diagnosed GBM patients is 14.6 months with a 2-year overall survival (OS) rate of 27.2%. This clinical trial evaluates the 2-year OS of oral NG101m as an adjuvant therapy to chemoradiotherapy in newly diagnosed GBM subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age
* Must be newly diagnosed with GBM
* Primary treatment must consist of a chemoradiation therapy (CRT) regimen
* Hemoglobin > 9 g/dL
* White blood count 3,600 - 11,000/mm3
* Absolute neutrophil count (ANC) ≥ 1,500/mm3
* Absolute lymphocyte count (ALC) ≥ 1,000/mm3
* Platelet count 100,000/mm3
* BUN ≤ 1.5 times upper limit of normal
* Creatinine clearance rate > 40 mL/min
* ALT ≤ 3 times upper limit of normal
* AST ≤ 3 times upper limit of normal
* Alkaline phosphatase ≤ 3 times upper limit of normal
* Total bilirubin ≤ 2.0 mg/dL
* Karnofsky Performance Status ≥ 70
* Must not be on any other alternative therapies
* Not pregnant

Exclusion Criteria:

* Known hypersensitivity to meloxicam, famotidine, and/or caffeine or any of their derivatives or components
* Known allergy to vitamin A, vitamin D3, and/or L-citrulline
* Pregnant women
* Breastfeeding women
* Corticosteroid therapy that cannot be tapered down to a dose of 1 - 2 mg/day of dexamethasone or its equivalent
* History of immunodeficiency diseases or autoimmune diseases
* History of peptic ulcer disease or gastrointestinal perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events and serious adverse events | 1 month
  Safety and tolerability of NG101m as adjuvant therapy to chemoradiation therapy
Efficacy of NG101m adjuvant chemoradiation therapy assessed by measuring 2-year overall survival rate. | 24 months
  Efficacy of NG101m adjuvant therapy will be assessed by measuring 2-year overall survival rate.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  Assess the duration of PFS
Response assessment in neuro-oncology (RANO) criteria | 24 months
  Radiological response to adjuvant NG101m therapy

OTHER OUTCOMES:
Identify and quantify immune/effector cells | 24 months
  Cytokines measurement

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Kew, MD, PhD, Study Director — NeuGATE Theranostics
Locations (1):
- Yvonne Kew MD, PLLC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No